CLINICAL TRIAL: NCT02017366
Title: Design of the EFECTS Trial, Investigating the Influence of Postoperative Enteral Feeding in Esophageal Cancer paTients on Survival
Brief Title: Design of the EFECTS Trial
Acronym: EFECTS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: adapted protocol with changed outcome measures, changed recruitment number, no submission to ethical board review
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Hans Van Veer, MD, MD, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EFECTS
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Cancer
Keywords: Surgery; Malnutrition; Nutrition, Enteral
MeSH Terms: conditions — Esophageal Neoplasms; Malnutrition | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group = standard of Care regimen: 1000ml = 1000 kCal TPN postop from day 1 until day 7. Oral feeds are started from day 5 onwards if no arguments for clinical leak (cervical anastomosis) or barium swallow is normal. Oral intake consists of regular post gastrectomy diet (building up from fluids over semi-solids to solids) with eventually added high nitrogen energy drinks.
- Enteral feeding (Active Comparator): Treatment group: start jejunostomy feeds from day 1, with target of 1000ml = 1000kCal (= 40cc/hour). To equilibrate energy intake during build up fase, Glucose 20% is given at a total cumulative dose taking into account the dose of j-drip, cumulative not exceeding 40cc/hr. Oral feeds are started at the same time as in the control group (reg. day 5) Jejunostomy feeds are then continued for 6 weeks together with oral intake with a continuous energy administration of 1000kCal, and then stopped. After this time, patients should be on regular full diet in both groups. If failure and step-back needed, temporary switch to Glc 20% is done to maintain fluid and calory administration.
  Interventions: Other: Enteral feeding

INTERVENTIONS:
Other: Enteral feeding — Target of 1000 kCal/day enteral feeding or glucose 20%, perferably given overnight.
  Arms: Enteral feeding

SUMMARY:
It is well known that there is a considerable postoperative weight loss in patients undergoing esophageal resection for cancer.

We believe that this weigh loss can be limited by administering postoperative enteral feeding (target: 1000 kCal/ day) via feeding jejunostomy for at least 6 weeks postoperatively.

We hypothesize that patients undergoing esophageal resection for cancer will have a better overall survival with postoperative additional enteral feeding than when on regular oral diet alone.

ELIGIBILITY:
Inclusion Criteria:

* advanced cT2 N+ or cT3 Nx
* all histology
* GEJ or distal esophageal ACC
* proximal or mid SCC
* curative intent with intention to treat
* no M+
* at least two-field lymphadenectomy
* all access: MIE, left thoraco freno or R thoraco + laparotomy with intrathoracic or cervical anastomosis
* all anastomosis (intrathoracic, cervical)

Exclusion Criteria:

* T4
* R2
* transhiatal
* pt in definitive CRT or rescue resection following definitive CRT
* palliative treatment
* tumours in cervical esophagus
* pharyngeal cancer with gastric pull-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
overall survival from day of surgery | 5 years postoperative
  overall survival at 5 years after esophagectomy

SECONDARY OUTCOMES:
postoperative weight loss | 1 year after surgery
  weight loss will be calculated by using age- and gender corrected BMI percentiles

CONTACTS AND LOCATIONS:
Overall Officials: Hans Van Veer, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Philippe Nafteux, MD, Study Chair — Universitaire Ziekenhuizen KU Leuven; Willy Coosemans, MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven; Johnny Moons, MScN, Study Chair — Universitaire Ziekenhuizen KU Leuven; Paul De Leyn, MD, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University hospital Leuven, Leuven, Vl-Brabant, Belgium